CLINICAL TRIAL: NCT05673109
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of AC176 in Chinese Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: A Study of AC176 for the Treatment of Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Subject benefit-risk ratio changes, sponsor decides to voluntarily terminate study
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC176-002
Record Dates: First submitted 2022-12-19; First posted 2023-01-06 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Metastatic Castration Resistant Prostate Cancer,; mCRPC;; Androgen Receptor,; Androgen Receptor Degrader,; AC176,; Phase 1
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC176 (Experimental): Single agent dose escalation of AC176. AC176 will be given orally (PO) on a 28-day cycle.
  Interventions: Drug: AC176

INTERVENTIONS:
Drug: AC176 — AC176 will be given orally (PO) on a 28-day cycle.

SUMMARY:
This clinical trial is evaluating a drug called AC176 in Chinese participants with metastatic castration resistant prostate cancer (mCRPC) who have progressed on at least one prior systemic therapy.

The main goals of this study are to:

Evaluate the safety and tolerability of AC176, evaluate pharmacokinetics and preliminary antitumor activity of AC176

DETAILED DESCRIPTION:
AC176-002 is a Phase I, open-label, multi-center dose-escalation study of AC176 given orally as a single agent. The AC176 is an investigational medicinal product that is a potent orally bioavailable Androgen Receptor (AR) degrader studied for the treatment of patients with metastatic castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients who are ≥ 18 years old when signing the ICF.
2. Patients with histologically, pathologically or cytologically confirmed mCRPC, except for any suspected neuroendocrine or small cell carcinoma. Patients with disease progression confirmed according to the Prostate Cancer Working Group 3 (PCWG3) Criteria, following standard of care, or for whom standard of care is inappropriate (they cannot tolerate or are unwilling to receive the standard of care), or for whom no therapy with proven efficacy is available.
3. Patients with disease progression meeting at least one of the following PCWG3 criteria:Positive bone scan (≥ 2 new lesions) or soft tissue metastases on CT/MRI ; or If PSA progression is the sole criterion for progression, its starting value of ≥ 1.0 ng/mL has been elevated twice at least 1 week apart.
4. Patients must have disease progression (in any stage of prostate cancer) after at least 1 of previously approved systemic therapies, at least 1 of which is Abiraterone, Enzalutamide, Apalutamide or Darolutamide.
5. The performance status score of the Eastern Cooperative Oncology Organization (ECOG) is 0-1.
6. Male patients with female partners of childbearing potential are required to use two forms of acceptable contraceptive measures.
7. Life expectancy ≥ 3 months after initiation of treatment, in the investigator's opinion.

Exclusion Criteria

Patients meeting any of the following criteria will be excluded from the study:

1. Patients who have received any of the following treatments:

   More than 2 lines of chemotherapy at any stage of prostate cancer treatment; Any systemic anti-cancer chemotherapy, biological agent in the previous treatment regimen or clinical study within 4 weeks prior to the first dose of the investigational drug; any systemic small molecule drug within 2 weeks prior to the first dose or 5 half-lives (whichever is longer, but no more than 4 weeks), except for the use of ADT for medical castration purposes; Any investigational drugs in previous clinical studies within 4 weeks before the first dose of the study treatment; Radiotherapy (including radioactive isotope therapy) within 4 weeks prior to the first dose of the investigational drug; or radiotherapy for remission within 2 weeks prior to the first dose. Palliative radiotherapy for relieving the pain caused by bone metastases.
2. Patients who have any > Grade 1 unresolved toxicity from prior therapy at the time of initiation of study treatment, except for alopecia and ≤ Grade 2 peripheral neuropathy (as assessed based on the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE]).
3. Patients who have received any major surgery(ies) (with the exception of the placement of vascular access) within 4 weeks prior to the first dose of the investigational drug.
4. Patients with known brain metastasis.
5. Male patients who plan to have children during the study or within 90 days after the last dose of investigational drug.
6. Patients who have any condition that impairs their ability to swallow a tablet whole, or have active gastrointestinal disease or other conditions that may significantly interfere with the absorption, distribution, metabolism or excretion of AC176
7. Patients whose cardiac functions currently meet or met the following criteria in the past 6 months:

   Mean corrected QT interval (QTc) in resting ECG is > 470 ms; Resting ECG shows clinically significant abnormalities ; Presence of any potential risk factors that may prolong QTc interval or increase the risk of arrhythmia, Left ventricular ejection fraction (LVEF) is < 50% or < the study site's LLN;
8. Patients presenting evidence(s) which is(are), in the opinion of the investigator, indicative of any serious or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses or active infection, with no need to screen for chronic diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs)/Serious adverse events (SAEs) | Through study completion, approximately 24 months
  Number of adverse events as characterized by type, frequency, seriousness, and relationship to AC176
Clinically significant abnormalities in vital signs | Through study completion, approximately 24 months
  Vital signs abnormalities as characterized by type, frequency, severity and timing;
Clinically significant abnormalities in laboratory tests | Through study completion, approximately 24 months
  Laboratory abnormalities as characterized by type, frequency, severity and timing;
Clinically significant abnormalities in electrocardiogram (ECG) | Through study completion, approximately 24 months
  Electrocardiogram (ECG) abnormalities such as QTcF, PR, RR and QRS intervals
Clinically significant abnormalities in heart rate | Through study completion, approximately 24 months

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) response rates based on Prostate Cancer Working Group 3 (PCWG3) criteria. | Throughout the study, approximately 24 months
  PSA response rate per PCWG3
Objective Response Rate(ORR) | Throughout the study, approximately 24 months
Radiographic progression-free survival (rPFS) | Throughout the study, approximately 24 months
Time to progression (TTP) | Throughout the study, approximately 24 months
Duration of response (DoR) | Throughout the study, approximately 24 months
Progression-free survival (PFS) | Throughout the study, approximately 24 months
Pharmacokinetic Analysis | 24 weeks
  Area under the concentration-time curve over the dosing interval (AUC(0-tau))
Pharmacokinetic Analysis | 24 weeks
  Maximum plasma concentration (Cmax)
Pharmacokinetic Analysis | 24 weeks
  Terminal elimination half life (t1/2)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Site 2001, Beijing
  - Site 2003, Guangzhou
  - Site 2004, Hunan
  - Site 2005, Nanchang
  - Site 2002, Shanghai

IPD SHARING:
Plan to Share IPD: No